CLINICAL TRIAL: NCT01877421
Title: A Double-Blind, Randomized, Controlled, Dose Escalation Clinical Trial of an Antiplaque Chewing Gum - Phase 1 Safety and Tolerability and Phase 2a Safety, Tolerability, and Proof of Concept in a Gingivitis Population
Brief Title: Safety and Tolerability of Antiplaque Chewing Gum in a Gingivitis Population
Acronym: APCG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-11-14
Record Dates: First submitted 2013-05-14; First posted 2013-06-13 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Plaque; Gingivitis
Keywords: Reducing plaque; Reducing gingivitis; safety; proof of concept; antiplaque chewing gum
MeSH Terms: conditions — Plaque, Amyloid; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- 2 mg KSL-W (Phase 1, 1a) (Experimental): one 2 mg KSL-W tablet at day 0 at Phase 1
  Interventions: Drug: 2 mg KSL-W
- 4 mg KSL-W (Phase 1, 2a; Phase 2a, 1b) (Experimental): one 4 mg KSL-W tablet on day 0 at both Phase 1 and Phase 2a. one 4 mg KSL-W tablet on days 1-6; two 4 mg KSL-W tablets on days 7-13 and days 14-20; and three 4 mg tablets at days 21-27 at Phase 2a.
  Interventions: Drug: 4 mg KSL-W
- 6 mg KSL-W (Phase 1, 3a; Phase 2a, 2b) (Experimental): One 6 mg KSL-W tablet on day 0 at both Phase 1 and Phase 2a. One 6 mg KSL-W tablet on days 1-6; two 6 mg KSL-W tablets on days 7-13 and days 14-20; and three 6 mg tablets at days 21-27 at Phase 2a.
  Interventions: Drug: 6 mg KSL-W
- 10 mg KSL-W (Phase 1, 4a; Phase 2a, 3b) (Experimental): One 10 mg KSL-W tablet on day 0 at both Phase 1 and Phase 2a. One 10 mg KSL-W tablet on days 1-6; two 10 mg KSL-W tablets on days 7-13 and days 14-20; and three 10 mg tablets at days 21-27 at Phase 2a.
  Interventions: Drug: 10 mg KSL-W
- 20 mg KSL-W (Phase 1, 5a; Phase 2a, 4b) (Experimental): One 20 mg KSL-W tablet on day 0 at both Phase 1 and Phase 2a. One 20 mg KSL-W tablet on days 1-6; two 20 mg KSL-W tablets on days 7-13 and days 14-20; and three 20 mg tablets at days 21-27 at Phase 2a.
  Interventions: Drug: 20 mg KSL-W
- 30 mg KSL-W (Phase 1, 6a; Phase 2a, 5b) (Experimental): One 30 mg KSL-W tablet on day 0 at both Phase 1 and Phase 2a. One 30 mg KSL-W tablet on days 1-6; two 30 mg KSL-W tablets on days 7-13 and days 14-20; and three 30 mg tablets at days 21-27 at Phase 2a.
  Interventions: Drug: 30 mg KSL-W
- 50 mg KSL-W (Phase 1, 7a; Phase 2a, 6b) (Experimental): One 50 mg KSL-W tablet on day 0 at both Phase 1 and Phase 2a. One 50 mg KSL-W tablet on days 1-6; two 50 mg KSL-W tablets on days 7-13 and days 14-20; and three 50 mg tablets at days 21-27 at Phase 2a.
  Interventions: Drug: 50 mg KSL-W
- 75 mg KSL-W (Phase 1, 8a; Phase 2a, 7b) (Experimental): One 75 mg KSL-W tablet on day 0 at both Phase 1 and Phase 2a. One 75 mg KSL-W tablet on days 1-6; two 75 mg KSL-W tablets on days 7-13 and days 14-20; and three 75 mg tablets at days 21-27 at Phase 2a.
  Interventions: Drug: 75 mg KSL-W
- 100 mg KSL-W (Phase 1, 9a) (Experimental): one 100 mg KSL-W tablet at day 0 at Phase 1
  Interventions: Drug: 100 mg KSL-W
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 2 mg KSL-W
  Other Names: Antiplaque Chewing Gum
  Arms: 2 mg KSL-W (Phase 1, 1a)
Drug: 4 mg KSL-W
  Other Names: Antiplaque Chewing Gum
  Arms: 4 mg KSL-W (Phase 1, 2a; Phase 2a, 1b)
Drug: 6 mg KSL-W
  Other Names: Antiplaque Chewing Gum
  Arms: 6 mg KSL-W (Phase 1, 3a; Phase 2a, 2b)
Drug: 10 mg KSL-W
  Other Names: Antiplaque Chewing Gum
  Arms: 10 mg KSL-W (Phase 1, 4a; Phase 2a, 3b)
Drug: 20 mg KSL-W
  Other Names: Antiplaque Chewing Gum
  Arms: 20 mg KSL-W (Phase 1, 5a; Phase 2a, 4b)
Drug: 30 mg KSL-W
  Other Names: Antiplaque Chewing Gum
  Arms: 30 mg KSL-W (Phase 1, 6a; Phase 2a, 5b)
Drug: 50 mg KSL-W
  Other Names: Antiplaque Chewing Gum
  Arms: 50 mg KSL-W (Phase 1, 7a; Phase 2a, 6b)
Drug: 75 mg KSL-W
  Other Names: Antiplaque Chewing Gum
  Arms: 75 mg KSL-W (Phase 1, 8a; Phase 2a, 7b)
Drug: 100 mg KSL-W
  Other Names: Antiplaque Chewing Gum
  Arms: 100 mg KSL-W (Phase 1, 9a)
Other: Placebo — Cetylpyridinium chloride (CPC) as an additive, isomalt as a bulk sweetener, peppermint powder for flavoring, sucralose as an intense sweetener, colloidal silicon dioxide is a flow enhancer, magnesium stearate as a process aid, and the proprietary gum base formulation.
  Arms: Placebo

SUMMARY:
This study is to assess the safety and tolerability of single doses and multiple doses in reducing plaque and gingivitis when delivered in a chewing gum formulation.

DETAILED DESCRIPTION:
This study is a Phase 1/2a placebo-controlled, double-blind, randomized, dose-escalation study to evaluate the safety and proof of concept of Antiplaque Chewing Gum. This is a 2-part trial with 9 dosing cohorts in Phase 1 and 7 dosing cohorts in Phase 2a. For both phases, the oral soft (OST) and oral hard tissues (OHT) will be examined. Changes from baseline, such as soft tissue erythema, ulceration and sloughing, will be noted and assessments will be made by the principal investigator as to whether they might be attributable to the antiplaque chewing gum.

In the Phase 2a portion of the study, the efficacy of the antiplaque chewing gum in reducing existing supragingival plaque and gingivitis will also be assessed. Plaque will be assessed using the Turesky Modification of the Quigley-Hein Plaque Index (PI, Turesky et al-1970) and gingivitis will be assessed using both the Modified Gingival Index (MGI, Lobene et al-1986) and the percent of bleeding sites on gentle probing (BOP) using the methods described in Ainamo and Bay-1975.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the Phase 1 portion of the study:

* Males and females between 18 and 64 years of age
* A negative urine pregnancy test and willingness to use a reliable form of contraception for the duration of the study (females of childbearing potential only), with reliable contraception defined as:

Abstinence Oral contraceptive, either estrogen progesterone combined, or progesterone alone Injectable progesterone Implants of levonorgestrel Estrogenic vaginal ring Percutaneous contraceptive patches Intrauterine device or intrauterine system Double barrier method [condom or occlusive cap (diaphragm or cervical vault caps) plus spermicidal agent (foam, gel, film, cream, suppository)] Male partner sterilization prior to the female subject's entry into the study, and this male is the sole partner for that subject

* Good health, as determined by pertinent medical history, physical examination, vital signs, and clinical safety laboratory evaluations
* A minimum of 16 natural teeth with 2 scorable surfaces (facial and lingual) per tooth Sufficient number of opposing posterior teeth to chew on both sides of the mouth as determined by the examining dentist Teeth that have gross caries, full crowns or extensive restorations on facial and/or lingual surfaces, orthodontic bands, and third molars are not included in the tooth count
* Ability to comprehend and a willingness to sign an informed consent, which includes the Authorization for the Release of Health Information document
* Willingness to comply with all study procedures

Phase 2a Inclusion Criteria

Subjects must meet all the criteria for the phase 1 portion of the study, and in addition must:

* Have mild to moderate gingivitis and plaque MGI of 1.8 or greater (Ainamo and Bay-1975) PI of 1.95 or greater (Turesky et al-1970)
* Willing to forgo any optional dental procedures during the study period, such as dental prophylaxis or teeth whitening

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

* Acute or chronic medical conditions, organ system disease, or medications that, in the principal investigator's opinion, would impair the subject's ability to participate
* TMD
* Self-reported use of tobacco products
* Use of anticoagulant medications (eg clopidogrel)
* Gross oral pathology, including widespread caries or chronic neglect, extensive restoration, pre-existing gross plaque or calculus, or soft or hard tissue tumor of the oral cavity
* Orthodontic appliances or removable partial dentures that will compromise the ability of the potential subject to participate in the study
* Periodontitis as indicated periodontal pockets greater than 4 millimeters on more than one site
* Receipt of any investigational drug/test product within 30 days prior to study entry
* Receipt of antibiotics within 30 days prior to study entry
* Need for antibiotic prophylaxis prior to invasive dental procedures
* Receipt of daily anti-inflammatory therapy [eg nonsteroidal anti-inflammatory drugs (NSAID), tumor necrosis factor (TNF) alpha blockers] within 30 days prior to study entry
* Receipt of prescription antibacterial oral products (eg products containing chlorhexidine) within 30 days prior to study entry
* Pregnant or breast-feeding female
* Clinically significant abnormal laboratory tests as determined by the principal investigator
* An employee of the study site directly involved with the study
* Inability to comply with assigned treatment regimen

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2015-08-25 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domenick T Zero, DDS, MS, Principal Investigator — Oral Health Research Institute, Indiana University School of Dentistry
Locations (1):
- Indiana University School of Dentistry, Oral Health Research Institute, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryan JB, Kirkwood BJ, Leung KP. Combined Phase 1/2a Initial Clinical Safety Trials and Proof-of-Concept Assessment of a Novel Antimicrobial Peptide KSL-W Anti-Plaque Chewing Gum. Clin Exp Dent Res. 2024 Dec;10(6):e943. doi: 10.1002/cre2.943. PMID 39466933

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were a total of 137 planned subjects (71 in Phase 1 and 66 in Phase 2) to participate in this study at the Oral Health Research Institute, Indiana University School of Dentistry. There were a total of 135 enrolled (71 in Phase 1 and 64 in Phase 2). Phase 1 and 2 are individual periods ran in parallel.
Groups:
- 2mg KSL-W: 2mg KSL-W
- 2mg Placebo: 2mg Placebo
- 4mg KSL-W: 4mg KSL-W
- 4mg Placebo: 4mg Placebo
- 6mg KSL-W: 6mg KSL-W
- 6mg Placebo: 6mg Placebo
- 10mg KSL-W: 10mg KSL-W
- 10mg Placebo: 10mg Placebo
- 20mg KSL-W: 20mg KSL-W
- 20mg Placebo: 20mg Placebo
- 30mg KSL-W: 30mg KSL-W
- 30mg Placebo: 30mg Placebo
- 50mg KSL-W: 50mg KSL-W
- 50mg Placebo: 50mg Placebo
- 75mg KSL-W: 75mg KSL-W
- 75mg Placebo: 75mg Placebo
- 100mg KSL-W: 100mg KSL-W
- 100mg Placebo: 100mg Placebo
Period: Phase 1
Arm/Group | 2mg KSL-W | 2mg Placebo | 4mg KSL-W | 4mg Placebo | 6mg KSL-W | 6mg Placebo | 10mg KSL-W | 10mg Placebo | 20mg KSL-W | 20mg Placebo | 30mg KSL-W | 30mg Placebo | 50mg KSL-W | 50mg Placebo | 75mg KSL-W | 75mg Placebo | 100mg KSL-W | 100mg Placebo
Started | 2 | 1 | 4 | 2 | 4 | 2 | 4 | 2 | 7 | 3 | 7 | 3 | 7 | 3 | 7 | 3 | 7 | 3
Completed | 2 | 1 | 4 | 2 | 4 | 2 | 4 | 2 | 7 | 3 | 7 | 3 | 7 | 3 | 7 | 3 | 7 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | 2mg KSL-W | 2mg Placebo | 4mg KSL-W | 4mg Placebo | 6mg KSL-W | 6mg Placebo | 10mg KSL-W | 10mg Placebo | 20mg KSL-W | 20mg Placebo | 30mg KSL-W | 30mg Placebo | 50mg KSL-W | 50mg Placebo | 75mg KSL-W | 75mg Placebo | 100mg KSL-W | 100mg Placebo
Started | 0 | 0 | 4 | 2 | 7 | 3 | 7 | 2 | 6 | 3 | 7 | 3 | 7 | 3 | 7 | 3 | 0 | 0
Completed | 0 | 0 | 4 | 2 | 7 | 3 | 6 | 2 | 5 | 3 | 5 | 3 | 6 | 3 | 7 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1, 1a (2mg): Subjects from phase 1, 1a (2mg) group
- Phase 1, 1a Placebo: Subjects from phase 1, 1a placebo group
- Phase 1, 2a (4mg); Phase 1, 2a Placebo: Subjects from phase 1, 2a (4mg) group
- Phase 1, 3a (6mg): Subject from phase 1, 3a (6mg) group
- Phase 1, 3a Placebo: Subjects from phase 1, 3a placebo gorup
- Phase 1, 4a (10mg): Subjects from phase 1, 4a (10mg) group
- Phase 1, 4a Placebo: Subjects from phase 1, 4a placebo group
- Phase 1, 5a (20mg): Subjects from phase 1, 5a (20mg) group
- Phase 1, 5a Placebo: Subjects from phase1, 5a placebo group
- Phase 1, 6a (30mg): Subjects from phase 1, 6a (30mg) group
- Phase 1, 6a Placebo: Subjects from phase 1, 6a placebo group
- Phase 1, 7a (50mg): Subjects from phase 1, 7a (50mg) group
- Phase 1, 7a Placebo: Subjects from phase 1, 7a placebo group
- Phase 1, 8a (75mg): Subjects from phase 1, 8a (75mg) group
- Phase 1, 8a Placebo: Subjects from phase 1, 8a placebo group
- Phase 1, 9a (100mg): Subjects from phase 1, 9a (100mg) group
- Phase 1, 9a Placebo: Subjects from phase 1, 9a placebo group
- Phase 2, 1b (4mg): Subjects from phase 2, 1b (4mg) group
- Phase 2, 1b Placebo: Subjects from phase 2, 1b placebo
- Phase 2, 2b (6mg): Subjects from phase 2, 2b (6mg) group
- Phase 2, 2b Placebo: Subjects from phase 2, 2b placebo group
- Phase 2, 3b (10mg): Subjects from phase 2, 3b (10mg) group
- Phase 2, 3b Placebo: Subjects from phase 2, 3b placebo group
- Phase 2, 4b (20mg): Subjects from phase 2, 4b (20mg) group
- Phase 2, 4b Placebo: Subjects from phase 2, 4b placebo group
- Phase 2, 5b (30mg): Subjects from phase 2, 5b (30mg) group
- Phase 2, 5b Placebo: Subjects from phase 2, 5b placebo group
- Phase 2, 6b (50mg): Subjects from phase 2, 6b (50mg) group
- Phase 2, 6b Placebo: Subjects from phase 2, 6b placebo group
- Phase 2, 7b (75mg): Subjects from phase 2, 7b (75mg) group
- Phase 2, 7b Placebo: Subjects from phase 2, 7b placebo group
- Total: Total of all reporting groups
Arm/Group | Phase 1, 1a (2mg) | Phase 1, 1a Placebo | Phase 1, 2a (4mg) | Phase 1, 2a Placebo | Phase 1, 3a (6mg) | Phase 1, 3a Placebo | Phase 1, 4a (10mg) | Phase 1, 4a Placebo | Phase 1, 5a (20mg) | Phase 1, 5a Placebo | Phase 1, 6a (30mg) | Phase 1, 6a Placebo | Phase 1, 7a (50mg) | Phase 1, 7a Placebo | Phase 1, 8a (75mg) | Phase 1, 8a Placebo | Phase 1, 9a (100mg) | Phase 1, 9a Placebo | Phase 2, 1b (4mg) | Phase 2, 1b Placebo | Phase 2, 2b (6mg) | Phase 2, 2b Placebo | Phase 2, 3b (10mg) | Phase 2, 3b Placebo | Phase 2, 4b (20mg) | Phase 2, 4b Placebo | Phase 2, 5b (30mg) | Phase 2, 5b Placebo | Phase 2, 6b (50mg) | Phase 2, 6b Placebo | Phase 2, 7b (75mg) | Phase 2, 7b Placebo | Total
Number analyzed (Participants) | 2 | 1 | 4 | 2 | 4 | 2 | 4 | 2 | 7 | 3 | 7 | 3 | 7 | 3 | 7 | 3 | 7 | 3 | 4 | 2 | 7 | 3 | 7 | 2 | 6 | 3 | 7 | 3 | 7 | 3 | 7 | 3 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (0.7) | 49.0 (NA) — SD not derived because n=1 | 31.8 (5.5) | 41.5 (2.1) | 29.8 (5.1) | 40.0 (5.7) | 44.5 (5.0) | 44.0 (11.3) | 38.0 (14.3) | 49.7 (9.5) | 36.7 (8.9) | 36.0 (5.6) | 27.4 (7.5) | 35.0 (19.1) | 29.3 (6.7) | 44.7 (13.6) | 26.4 (10.4) | 33.7 (20.6) | 31.5 (11.4) | 36.5 (16.3) | 38.1 (12.2) | 22.0 (3.6) | 25.7 (5.8) | 33.0 (15.6) | 30.2 (14.3) | 34.3 (13.6) | 21.3 (4.8) | 24.0 (5.0) | 37.3 (13.9) | 26.0 (10.4) | 26.0 (5.0) | 21.7 (0.6) | 21.3 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 1 | 2 | 0 | 0 | 1 | 4 | 1 | 5 | 3 | 6 | 3 | 5 | 3 | 5 | 2 | 1 | 0 | 5 | 1 | 1 | 1 | 3 | 1 | 2 | 2 | 5 | 2 | 3 | 2 | 76
  Male | 0 | 0 | 1 | 1 | 2 | 2 | 4 | 1 | 3 | 2 | 2 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 3 | 2 | 2 | 2 | 6 | 1 | 3 | 2 | 5 | 1 | 2 | 1 | 4 | 1 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 13
  Not Hispanic or Latino | 2 | 1 | 4 | 2 | 3 | 2 | 4 | 2 | 3 | 3 | 6 | 3 | 7 | 3 | 7 | 2 | 4 | 2 | 3 | 2 | 7 | 3 | 7 | 2 | 6 | 3 | 7 | 3 | 7 | 3 | 6 | 3 | 122
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 0 | 22
  White | 0 | 1 | 3 | 2 | 4 | 2 | 3 | 1 | 7 | 2 | 5 | 3 | 5 | 3 | 6 | 2 | 4 | 1 | 2 | 2 | 4 | 1 | 4 | 1 | 6 | 3 | 4 | 2 | 6 | 2 | 2 | 2 | 95
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 4 | 2 | 4 | 2 | 4 | 2 | 7 | 3 | 7 | 3 | 7 | 3 | 7 | 3 | 7 | 3 | 4 | 2 | 7 | 3 | 7 | 2 | 6 | 3 | 7 | 3 | 7 | 3 | 7 | 3 | 135

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of KSL-W as Measured by Soft Tissue Erythema, Ulceration and Sloughing (AEs and SAEs)
Description: Occurrence of local oral mucosal reactions, systemic reactions such as fever, nausea, headache, and changes in blood pressure, clinical laboratory measures of safety, and serious total body reactions will be assessed (AEs and SAEs)
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, 1a (2mg) | Phase 1, 1a Placebo | Phase 1, 2a (4mg) | Phase 1, 2a Placebo | Phase 1, 3a (6mg) | Phase 1, 3a Placebo | Phase 1, 4a (10mg) | Phase 1, 4a Placebo | Phase 1, 5a (20mg) | Phase 1, 5a Placebo | Phase 1, 6a (30mg) | Phase 1, 6a Placebo | Phase 1, 7a (50mg) | Phase 1, 7a Placebo | Phase 1, 8a (75mg) | Phase 1, 8a Placebo | Phase 1, 9a (100mg) | Phase 1, 9a Placebo | Phase 2, 1b (4mg) | Phase 2, 1b Placebo | Phase 2, 2b (6mg) | Phase 2, 2b Placebo | Phase 2, 3b (10mg) | Phase 2, 3b Placebo | Phase 2, 4b (20mg) | Phase 2, 4b Placebo | Phase 2, 5b (30mg) | Phase 2, 5b Placebo | Phase 2, 6b (50mg) | Phase 2, 6b Placebo | Phase 2, 7b (75mg) | Phase 2, 7b Placebo
Number analyzed (Participants) | 2 | 1 | 4 | 2 | 4 | 2 | 4 | 2 | 7 | 3 | 7 | 3 | 7 | 3 | 7 | 3 | 7 | 3 | 4 | 2 | 7 | 3 | 7 | 2 | 6 | 3 | 7 | 3 | 7 | 3 | 7 | 3
Participants
  Subject Experiencing AEs = NO | 2 | 1 | 4 | 2 | 4 | 1 | 4 | 1 | 6 | 1 | 7 | 3 | 7 | 3 | 5 | 3 | 5 | 3 | 2 | 1 | 4 | 2 | 4 | 2 | 5 | 1 | 2 | 1 | 2 | 2 | 2 | 3
  Subjects Experiencing AEs = YES | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 1 | 3 | 1 | 3 | 0 | 1 | 2 | 5 | 2 | 5 | 1 | 5 | 0

2. Secondary Outcome: Proof of Concept of KSL-W in Reducing Plaque in Phase 2a
Description: Data summarizes plaque index scores changes from baseline. Supragingival plaque will be assessed after the MGI and BOP assessments and following use of a disclosing solution on the facial (buccal) and lingual surfaces of a minimum of 16 scorable teeth according to the criteria of the Turesky modification of the Quigley-Hein Plaque Index.
  Quigley-Hein Plaque Index Scores with Turesky Modifications:
  0 No plaque
  1. Separate flecks of plaque at the cervical margin of the tooth
  2. A thin continuous band of plaque (up to one mm) at the cervical margin of the tooth
  3. A band of plaque wider than one mm but covering less than one-third of the crown of the tooth
  4. Plaque covering at least one-third but less than two thirds of the crown of the tooth
  5. Plaque covering two-thirds or more of the crown of the tooth
Time Frame: days 14, 28, 34
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Phase 2, 1b (4mg) | Phase 2, 1b Placebo | Phase 2, 2b (6mg) | Phase 2, 2b Placebo | Phase 2, 3b (10mg) | Phase 2, 3b Placebo | Phase 2, 4b (20mg) | Phase 2, 4b Placebo | Phase 2, 5b (30mg) | Phase 2, 5b Placebo | Phase 2, 6b (50mg) | Phase 2, 6b Placebo | Phase 2, 7b (75mg) | Phase 2, 7b Placebo
Number analyzed (Participants) | 4 | 2 | 7 | 3 | 7 | 2 | 5 | 3 | 6 | 3 | 7 | 3 | 7 | 3
scores on a scale
  Whole Mouth: Day 14 | 0.20 (0.30) | -0.06 (0.02) | -0.12 (0.16) | -0.10 (0.39) | 0.01 (0.15) | 0.04 (0.10) | -0.08 (0.15) | 0.01 (0.12) | -0.31 (0.23) | -0.14 (0.08) | -0.52 (0.25) | 0.06 (0.12) | -0.53 (0.44) | 0.28 (0.12)
  Whole Mouth: Day 28 | 0.37 (0.42) | -0.11 (0.07) | -0.19 (0.10) | 0.03 (0.08) | 0.19 (0.21) | 0.10 (0.10) | -0.20 (0.09) | 0.02 (0.15) | -0.40 (0.36) | -0.05 (0.03) | -0.42 (0.20) | 0.05 (0.15) | -0.59 (0.54) | 0.22 (0.11)
  Whole Mouth: Day 34 | 0.22 (0.24) | 0.00 (0.07) | -0.17 (0.23) | -0.16 (0.43) | 0.25 (0.26) | -0.01 (0.06) | -0.08 (0.02) | 0.00 (0.10) | -0.21 (0.26) | -0.04 (0.10) | -0.18 (0.33) | -0.17 (0.24) | -0.20 (0.44) | 0.49 (0.32)
  Maxillary: Day 14 | 0.21 (0.44) | -0.01 (0.11) | -0.17 (0.21) | -0.17 (0.40) | -0.02 (0.21) | -0.01 (0.14) | -0.07 (0.24) | 0.01 (0.15) | -0.35 (0.31) | -0.11 (0.09) | -0.53 (0.27) | 0.06 (0.10) | -0.59 (0.52) | 0.36 (0.03)
  Maxillary: Day 28 | 0.41 (0.51) | 0.03 (0.13) | -0.19 (0.10) | 0.01 (0.12) | 0.13 (0.24) | 0.06 (0.15) | -0.22 (0.16) | 0.08 (0.19) | -0.49 (0.43) | -0.03 (0.08) | -0.38 (0.28) | 0.06 (0.15) | -0.56 (0.56) | 0.24 (0.09)
  Maxillary: Day 34 | 0.21 (0.31) | 0.02 (0.19) | -0.23 (0.20) | -0.16 (0.32) | 0.24 (0.25) | -0.02 (0.01) | -0.04 (0.07) | 0.04 (0.12) | -0.18 (0.35) | -0.01 (0.13) | -0.25 (0.34) | -0.21 (0.26) | -0.23 (0.50) | 0.68 (0.31)
  Mandibular: Day 14 | 0.19 (0.19) | -0.13 (0.07) | -0.07 (0.17) | -0.02 (0.38) | 0.014 (0.16) | 0.09 (0.06) | -0.09 (0.14) | 0.00 (0.08) | -0.27 (0.19) | -0.17 (0.058) | -0.50 (0.26) | 0.06 (0.14) | -0.48 (0.38) | 0.20 (0.23)
  Mandibular: Day 28 | 0.33 (0.36) | -0.26 (0.27) | -0.20 (0.21) | 0.06 (0.06) | 0.24 (0.21) | 0.13 (0.05) | -0.19 (0.05) | -0.05 (0.24) | -0.31 (0.31) | -0.07 (0.07) | -0.46 (0.20) | 0.04 (0.17) | -0.62 (0.53) | 0.19 (0.12)
  Mandibular: Day 34 | 0.24 (0.174) | -0.03 (0.05) | -0.11 (0.28) | -0.16 (0.54) | 0.26 (0.30) | 0.00 (0.12) | -0.11 (0.04) | -0.04 (0.15) | -0.23 (0.18) | -0.07 (0.12) | -0.12 (0.32) | -0.14 (0.22) | -0.17 (0.38) | 0.30 (0.32)
  Posterior: Day 14 | 0.14 (0.26) | -0.04 (0.09) | -0.20 (0.22) | 0.08 (0.16) | -0.06 (0.15) | 0.00 (0.31) | -0.10 (0.14) | 0.09 (0.07) | -0.45 (0.33) | -0.22 (0.14) | -0.66 (0.30) | 0.04 (0.18) | -0.60 (0.44) | 0.31 (0.17)
  Posterior: Day 28 | 0.39 (0.34) | -0.18 (0.05) | -0.30 (0.13) | 0.08 (0.06) | 0.09 (0.20) | 0.05 (0.15) | -0.25 (0.10) | 0.03 (0.21) | -0.58 (0.44) | -0.14 (0.14) | -0.52 (0.19) | 0.04 (0.16) | -0.69 (0.54) | 0.22 (0.16)
  Posterior: Day 34 | 0.27 (0.15) | 0.00 (0.09) | -0.24 (0.22) | 0.08 (0.23) | 0.24 (0.24) | -0.03 (0.10) | -0.10 (0.07) | 0.06 (0.19) | -1.31 (0.31) | -0.07 (0.15) | -0.18 (0.39) | -0.21 (0.37) | -0.18 (0.40) | 0.53 (0.37)
  Interproximal: Day 14 | 0.25 (0.31) | 0.02 (0.15) | -0.12 (0.24) | -0.10 (0.36) | 0.09 (0.19) | 0.06 (0.04) | -0.08 (0.11) | 0.03 (0.08) | -0.36 (0.33) | -0.20 (0.08) | 0.61 (0.29) | 0.04 (0.18) | -0.58 (0.49) | 0.32 (0.08)
  Interproximal: Day 28 | 0.41 (0.46) | -0.08 (0.06) | -0.20 (0.13) | -0.03 (0.07) | 0.28 (0.28) | 0.12 (0.05) | -0.22 (0.12) | -0.02 (0.09) | -0.60 (0.39) | -0.21 (0.07) | -0.53 (0.25) | 0.02 (0.10) | -0.67 (0.61) | 0.24 (0.20)
  Interproximal: Day 34 | 0.30 (0.21) | 0.06 (0.08) | -0.18 (0.27) | -0.16 (0.41) | 0.37 (0.34) | -0.01 (0.12) | -0.07 (0.05) | -0.06 (0.03) | -0.24 (0.28) | -0.05 (0.11) | -0.24 (0.43) | -0.21 (0.24) | -0.18 (0.44) | 0.54 (0.40)
  Facial: Day 14 | 0.30 (0.47) | -0.17 (0.04) | -0.08 (0.24) | -0.09 (0.47) | 0.07 (0.18) | 0.03 (0.16) | -0.06 (0.17) | -0.02 (0.19) | -0.20 (0.28) | -0.06 (0.21) | -0.45 (0.37) | 0.10 (0.03) | -0.60 (0.55) | 0.31 (0.17)
  Facial: Day 28 | 0.52 (0.65) | -0.20 (0.03) | -0.18 (0.20) | 0.11 (0.10) | 0.24 (0.29) | 0.02 (0.13) | -0.08 (0.10) | 0.06 (0.21) | -0.16 (0.43) | 0.07 (0.14) | -0.37 (0.36) | -0.03 (0.23) | -0.70 (0.69) | 0.29 (0.20)
  Facial: Day 34 | 0.25 (0.44) | -0.14 (0.16) | -0.12 (0.29) | -0.16 (0.54) | 0.28 (0.40) | -0.12 (0.04) | -0.05 (0.08) | 0.03 (0.08) | -0.08 (0.41) | -0.04 (0.09) | -0.17 (0.36) | -0.22 (0.29) | -0.25 (0.60) | 0.57 (0.35)
  Lingual: Day 14 | 0.10 (0.14) | 0.04 (0.09) | -0.16 (0.19) | 0.11 (0.31) | -0.05 (0.15) | 0.06 (0.04) | -0.10 (0.21) | 0.03 (0.05) | -0.43 (0.26) | -0.22 (0.10) | -0.59 (0.23) | 0.03 (0.21) | -0.47 (0.41) | 0.25 (0.08)
  Lingual: Day 28 | 0.22 (0.24) | -0.02 (0.10) | -0.20 (0.19) | -0.06 (0.11) | 0.14 (0.23) | 0.17 (0.07) | -0.32 (0.18) | -0.02 (0.11) | -0.64 (0.41) | -0.16 (0.17) | -0.47 (0.17) | 0.13 (0.10) | -0.48 (0.40) | 0.15 (0.01)
  Lingual: Day 34 | 0.20 (0.08) | 0.14 (0.02) | -0.22 (0.28) | -0.16 (0.32) | 0.22 (0.26) | 0.10 (0.08) | -0.11 (0.11) | -0.02 (0.12) | -0.33 (0.13) | -0.03 (0.16) | -0.20 (0.34) | -0.12 (0.18) | -0.14 (0.32) | 0.42 (0.29)

3. Secondary Outcome: Proof of Concept of KSL-W in Reducing Gingivitis in Phase 2a
Description: Data summarizes gingival index scores changes from baseline in phase 2a. Gingivitis will be assessed using both the MGI (Modified Gingival Index) and the Gingival Bleeding Index (BOP) The Modified Gingival Index assesses the buccal and lingual gingivae and interdental papillae.
  Modified Gingival Index Scores:
  0 Absence of inflammation
  1. Mild inflammation; slight change in color, little change in texture of any portion of but not the entire marginal or papillary gingival unit
  2. Mild inflammation; criteria as above but involving the entire marginal or papillary gingival unit
  3. Moderate inflammation; glazing, redness, edema and/or hypertrophy of the marginal or papillary gingival unit
  4. Severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration.
Time Frame: days 14, 28, 34
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Phase 2, 1b (4mg) | Phase 2, 1b Placebo | Phase 2, 2b (6mg) | Phase 2, 2b Placebo | Phase 2, 3b (10mg) | Phase 2, 3b Placebo | Phase 2, 4b (20mg) | Phase 2, 4b Placebo | Phase 2, 5b (30mg) | Phase 2, 5b Placebo | Phase 2, 6b (50mg) | Phase 2, 6b Placebo | Phase 2, 7b (75mg) | Phase 2, 7b Placebo
Number analyzed (Participants) | 4 | 2 | 7 | 3 | 7 | 2 | 5 | 3 | 6 | 3 | 7 | 3 | 7 | 3
scores on a scale
  Whole Mouth: Day 14 | -0.03 (0.05) | -0.06 (0.09) | 0.00 (0.04) | 0.14 (0.10) | 0.04 (0.11) | 0.10 (0.04) | 0.01 (0.03) | 0.05 (0.03) | -0.11 (0.08) | -0.12 (0.09) | -0.03 (0.12) | 0.00 (0.18) | -0.10 (0.11) | 0.00 (0.07)
  Whole Mouth: Day 28 | 0.10 (0.06) | 0.04 (0.02) | 0.00 (0.07) | 0.06 (0.10) | 0.03 (0.12) | 0.14 (0.07) | 0.07 (0.03) | 0.08 (0.13) | -0.13 (0.06) | -0.09 (0.13) | -0.02 (0.09) | -0.11 (0.11) | -0.10 (0.08) | 0.12 (0.10)
  Whole Mouth: Day 34 | 0.05 (0.10) | 0.02 (0.08) | -0.01 (0.09) | 0.06 (0.04) | -0.05 (0.08) | 0.02 (0.08) | 0.04 (0.04) | -0.03 (0.09) | -0.15 (0.04) | 0.13 (0.08) | -0.04 (0.07) | -0.08 (0.09) | -0.05 (0.08) | 0.16 (0.00)
  Maxillary: Day 14 | -0.06 (0.03) | -0.08 (0.10) | 0.01 (0.10) | 0.15 (0.13) | 0.02 (0.14) | 0.11 (0.05) | 0.00 (0.09) | -0.02 (0.05) | -0.11 (0.08) | -0.05 (0.08) | -0.03 (0.19) | -0.04 (0.25) | -0.17 (0.11) | 0.02 (0.04)
  Maxillary: Day 28 | 0.01 (0.06) | 0.04 (0.07) | 0.00 (0.14) | 0.01 (0.19) | 0.06 (0.17) | 0.09 (0.09) | 0.08 (0.05) | 0.03 (0.19) | -0.12 (0.07) | -0.03 (0.18) | 0.00 (0.11) | -0.15 (0.16) | -0.12 (0.09) | 0.15 (0.06)
  Maxillary: Day 34 | -0.02 (0.12) | 0.00 (0.07) | -0.02 (0.15) | 0.01 (0.16) | -0.03 (0.16) | -0.02 (0.06) | 0.01 (0.09) | -0.09 (0.14) | -0.15 (0.08) | -0.09 (0.11) | -0.06 (0.05) | -0.12 (0.09) | -0.12 (0.08) | 0.16 (0.09)
  Mandibular: Day 14 | 0.00 (0.09) | -0.03 (0.09) | 0.00 (0.08) | 0.12 (0.18) | 0.07 (0.09) | 0.10 (0.03) | 0.01 (0.05) | 0.13 (0.07) | -0.10 (0.10) | -0.19 (0.11) | -0.02 (0.07) | 0.03 (0.10) | -0.02 (0.13) | -0.02 (0.12)
  Mandibular: Day 28 | 0.18 (0.08) | 0.05 (0.03) | -0.01 (0.11) | 0.11 (0.06) | 0.00 (0.08) | 0.19 (0.05) | 0.05 (0.05) | 0.12 (0.07) | -0.14 (0.06) | -0.15 (0.07) | -0.04 (0.12) | -0.07 (0.10) | -0.07 (0.09) | 0.10 (0.13)
  Mandibular: Day 34 | 0.13 (0.09) | 0.05 (0.08) | 0.01 (0.047) | 0.10 (0.09) | -0.06 (0.07) | 0.07 (0.11) | 0.07 (0.06) | 0.03 (0.08) | -0.14 (0.11) | -0.17 (0.07) | -0.01 (0.13) | -0.04 (0.12) | 0.01 (0.10) | 0.17 (0.08)
  Posterior: Day 14 | 0.00 (0.04) | -0.05 (0.07) | 0.00 (0.11) | 0.10 (0.11) | 0.05 (0.11) | 0.11 (0.10) | -0.01 (0.02) | 0.03 (0.04) | -0.11 (0.12) | -0.10 (0.15) | 0.00 (0.11) | 0.01 (0.14) | -0.11 (0.10) | 0.00 (0.05)
  Posterior: Day 28 | 0.17 (0.10) | 0.02 (0.02) | 0.01 (0.07) | 0.06 (0.11) | 0.02 (0.11) | 0.19 (0.07) | 0.12 (0.05) | 0.10 (0.08) | -0.10 (0.06) | -0.12 (0.19) | 0.04 (0.10) | -0.12 (0.14) | -0.11 (0.10) | 0.08 (0.05)
  Posterior: Day 34 | 0.06 (0.09) | 0.09 (0.01) | -0.02 (0.14) | 0.06 (0.04) | -0.03 (0.06) | 0.08 (0.15) | 0.06 (0.05) | -0.04 (0.07) | -0.13 (0.11) | -0.14 (0.14) | -0.03 (0.07) | -0.09 (0.05) | -0.08 (0.06) | 0.15 (0.01)
  Interproximal: Day 14 | -0.03 (0.05) | -0.06 (0.09) | 0.02 (0.06) | 0.12 (0.11) | 0.04 (0.10) | 0.09 (0.01) | 0.00 (0.02) | 0.08 (0.08) | -0.10 (0.10) | -0.08 (0.08) | -0.01 (0.13) | -0.01 (0.19) | -0.11 (0.13) | -0.06 (0.07)
  Interproximal: Day 28 | 0.02 (0.06) | 0.01 (0.06) | 0.03 (0.03) | 0.05 (0.08) | 0.04 (0.10) | 0.16 (0.03) | 0.07 (0.06) | 0.10 (0.11) | -0.14 (0.06) | -0.05 (0.13) | 0.01 (0.08) | -0.10 (0.15) | -0.11 (0.09) | 0.08 (0.14)
  Interproximal: Day 34 | 0.02 (0.11) | 0.02 (0.04) | 0.01 (0.08) | 0.05 (0.02) | -0.06 (0.07) | 0.01 (0.09) | 0.03 (0.05) | 0.00 (0.12) | -0.15 (0.05) | -0.09 (0.05) | -0.02 (0.07) | -0.08 (0.10) | -0.07 (0.09) | 0.18 (0.03)
  Facial: Day 14 | 0.04 (0.10) | -0.05 (0.14) | -0.04 (0.11) | 0.10 (0.09) | 0.02 (0.13) | 0.05 (0.08) | 0.00 (0.03) | 0.05 (0.09) | -0.08 (0.05) | -0.09 (0.14) | -0.06 (0.15) | 0.04 (0.22) | -0.05 (0.09) | -0.05 (0.08)
  Facial: Day 28 | 0.19 (0.14) | 0.02 (0.03) | 0.00 (0.09) | 0.08 (0.08) | 0.01 (0.13) | 0.16 (0.04) | 0.09 (0.09) | 0.10 (0.00) | -0.11 (0.08) | -0.06 (0.17) | -0.05 (0.12) | -0.11 (0.15) | -0.07 (0.06) | 0.09 (0.08)
  Facial: Day 34 | 0.09 (0.16) | -0.05 (0.09) | -0.02 (0.15) | 0.10 (0.047) | -0.04 (0.08) | -0.05 (0.02) | 0.01 (0.07) | -0.07 (0.14) | -0.12 (0.03) | -0.10 (0.09) | -0.06 (0.09) | -0.09 (0.12) | -0.04 (0.07) | 0.19 (0.00)
  Lingual: Day 14 | -0.10 (0.10) | -0.06 (0.05) | 0.05 (0.10) | 0.18 (0.12) | 0.06 (0.14) | 0.15 (0.15) | 0.01 (0.06) | 0.06 (0.07) | -0.13 (0.13) | -0.15 (0.04) | 0.00 (0.10) | -0.05 (0.14) | -0.14 (0.16) | 0.05 (0.07)
  Lingual: Day 28 | 0.00 (0.09) | 0.07 (0.01) | 0.00 (0.07) | 0.03 (0.13) | 0.05 (0.14) | 0.12 (0.19) | 0.05 (0.08) | 0.06 (0.25) | -0.15 (0.06) | -0.12 (0.08) | 0.01 (0.10) | -0.12 (0.08) | -0.13 (0.11) | 0.15 (0.12)
  Lingual: Day 34 | 0.01 (0.07) | 0.10 (0.07) | 0.00 (0.09) | 0.02 (0.16) | -0.05 (0.14) | 0.10 (0.15) | 0.08 (0.06) | 0.01 (0.04) | -0.17 (0.07) | -0.17 (0.08) | -0.01 (0.07) | -0.07 (0.07) | -0.06 (0.14) | 0.14 (0.01)

4. Secondary Outcome: Gingival Bleeding on Probing (BOP) - Percent of Bleeding Sites Upon Probing in Phase 2a
Description: Proof of concept of KSL-W in reducing plaque as measured by percent of bleeding sites upon probing (BOP) in phase 2a.
  Gingivitis will be assessed using both the MGI (Modified Gingival Index) and the Gingival Bleeding Index (BOP). The Modified Gingival Index assesses the buccal and lingual gingivae and interdental papillae. The Gingival Bleeding Index assesses the percentage of sites that bleed on gentle probing. A periodontal probe (HU-Friedy UNC 15) will be gently inserted into the gingival sulcus until resistance is felt at mid-facial (buccal), mid-lingual, mesial, and distal interproximal sites of all scorable teeth, with the exception of the most posterior distal sites. Presence or absence of bleeding will be recorded for each site and the percentage of bleeding sites per subject will serve as the unit of analysis.
Time Frame: days 0, 14, 28, 34
Measure: Mean (Standard Deviation); unit: Percent of bleeding sites
Arm/Group | Phase 2, 1b (4mg) | Phase 2, 1b Placebo | Phase 2, 2b (6mg) | Phase 2, 2b Placebo | Phase 2, 3b (10mg) | Phase 2, 3b Placebo | Phase 2, 4b (20mg) | Phase 2, 4b Placebo | Phase 2, 5b (30mg) | Phase 2, 5b Placebo | Phase 2, 6b (50mg) | Phase 2, 6b Placebo | Phase 2, 7b (75mg) | Phase 2, 7b Placebo
Number analyzed (Participants) | 4 | 2 | 7 | 3 | 7 | 2 | 6 | 3 | 7 | 3 | 7 | 3 | 7 | 3
Percent of bleeding sites
  Whole Mouth: Eligibility | 16 (15) | 27 (26) | 26 (10) | 22 (16) | 17 (16) | 27 (7) | 30 (14) | 37 (26) | 25 (8) | 17 (5) | 20 (15) | 19 (8) | 13 (9) | 11 (9)
  Whole Mouth: Day 0 | 20 (12) | 37 (31) | 29 (12) | 19 (6) | 16 (11) | 26 (5) | 29 (19) | 38 (28) | 31 (14) | 19 (8) | 25 (19) | 27 (12) | 21 (16) | 17 (4)
  Whole Mouth: Day 14 | 16 (15) | 28 (24) | 21 (11) | 24 (13) | 17 (15) | 15 (11) | 25 (17) | 33 (20) | 24 (14) | 20 (14) | 19 (8) | 32 (1) | 15 (7) | 15 (9)
  Whole Mouth: Day 28 | 16 (18) | 24 (29) | 25 (9) | 23 (14) | 13 (10) | 25 (12) | 33 (21) | 28 (8) | 25 (16) | 24 (3) | 17 (17) | 31 (18) | 22 (9) | 13 (1)
  Whole Mouth: Day 34 | 18 (18) | 46 (11) | 18 (10) | 22 (15) | 16 (12) | 28 (27) | 31 (17) | 31 (21) | 22 (13) | 12 (6) | 10 (5) | 24 (14) | 19 (10) | 20 (4)
  Maxillary: Eligibility | 16 (18) | 26 (25) | 26 (11) | 29 (15) | 17 (15) | 29 (14) | 33 (20) | 37 (22) | 26 (12) | 17 (8) | 23 (20) | 16 (3) | 14 (8) | 8 (5)
  Maxillary: Day 0 | 24 (19) | 30 (29) | 27 (11) | 21 (3) | 17 (12) | 21 (2) | 31 (28) | 37 (23) | 29 (13) | 20 (11) | 32 (24) | 22 (11) | 22 (17) | 20 (6)
  Maxillary: Day 14 | 19 (25) | 30 (29) | 21 (16) | 33 (15) | 19 (16) | 12 (2) | 29 (21) | 33 (15) | 26 (17) | 16 (12) | 24 (12) | 36 (7) | 14 (12) | 15 (6)
  Maxillary: Day 28 | 14 (14) | 26 (29) | 25 (10) | 27 (17) | 15 (13) | 21 (14) | 31 (23) | 30 (10) | 231 (16) | 26 (5) | 18 (17) | 30 (21) | 24 (12) | 15 (4)
  Maxillary: Day 34 | 22 (26) | 39 (11) | 19 (13) | 25 (15) | 15 (10) | 26 (27) | 28 (18) | 29 (17) | 22 (13) | 13 (10) | 11 (3) | 24 (14) | 18 (9) | 17 (2)
  Mandibular: Eligibility | 16 (12) | 28 (28) | 26 (12) | 15 (18) | 17 (18) | 26 (1) | 27 (12) | 36 (30) | 24 (7) | 17 (5) | 16 (12) | 22 (14) | 11 (11) | 15 (13)
  Mandibular: Day 0 | 17 (6) | 43 (32) | 31 (15) | 18 (14) | 15 (11) | 32 (8) | 26 (13) | 39 (34) | 32 (17) | 17 (7) | 18 (14) | 33 (16) | 20 (17) | 13 (3)
  Mandibular: Day 14 | 13 (8) | 27 (19) | 20 (10) | 16 (13) | 16 (15) | 18 (21) | 21 (14) | 34 (28) | 22 (15) | 25 (17) | 15 (6) | 28 (6) | 17 (12) | 15 (12)
  Mandibular: Day 28 | 17 (22) | 23 (29) | 25 (12) | 19 (12) | 12 (9) | 29 (10) | 34 (20) | 27 (8) | 28 (17) | 22 (2) | 17 (17) | 32 (17) | 19 (12) | 11 (3)
  Mandibular: Day 34 | 15 (11) | 52 (10) | 17 (10) | 18 (16) | 16 (15) | 30 (26) | 34 (18) | 34 (26) | 22 (15) | 10 (4) | 9 (12) | 25 (14) | 21 (15) | 23 (9)
  Posterior: Eligibility | 21 (21) | 24 (23) | 30 (12) | 28 (10) | 21 (19) | 29 (13) | 34 (16) | 36 (17) | 25 (9) | 19 (6) | 22 (16) | 21 (10) | 14 (11) | 12 (6)
  Posterior: Day 0 | 25 (11) | 40 (32) | 32 (15) | 22 (5) | 20 (13) | 33 (5) | 30 (19) | 38 (25) | 32 (15) | 20 (6) | 27 (21) | 34 (16) | 24 (21) | 19 (7)
  Posterior: Day 14 | 19 (20) | 32 (26) | 26 (15) | 34 (9) | 23 (19) | 17 (7) | 28 (16) | 35 (17) | 27 (14) | 19 (9) | 23 (9) | 39 (3) | 17 (7) | 16 (12)
  Posterior: Day 28 | 20 (24) | 26 (29) | 29 (9) | 30 (17) | 17 (14) | 30 (21) | 34 (22) | 30 (10) | 24 (15) | 27 (4) | 20 (19) | 34 (20) | 24 (10) | 14 (0)
  Posterior: Day 34 | 22 (21) | 45 (18) | 23 (9) | 26 (10) | 19 (14) | 31 (32) | 32 (16) | 33 (21) | 24 (14) | 13 (6) | 13 (5) | 27 (13) | 20 (12) | 27 (7)
  Interproximal: Eligibility | 21 (19) | 32 (32) | 32 (12) | 30 (23) | 20 (19) | 38 (9) | 37 (18) | 44 (29) | 30 (9) | 21 (4) | 24 (18) | 22 (8) | 16 (10) | 14 (10)
  Interproximal: Day 0 | 25 (14) | 39 (28) | 36 (15) | 24 (8) | 19 (13) | 34 (4) | 34 (21) | 45 (33) | 36 (17) | 21 (8) | 29 (20) | 33 (15) | 24 (19) | 20 (7)
  Interproximal: Day 14 | 20 (20) | 34 (26) | 26 (14) | 32 (17) | 20 (18) | 20 (14) | 31 (22) | 39 (23) | 28 (17) | 25 (22) | 23 (11) | 36 (3) | 17 (8) | 17 (11)
  Interproximal: Day 28 | 19 (21) | 29 (32) | 32 (11) | 31 (20) | 16 (11) | 30 (13) | 38 (26) | 35 (8) | 26 (16) | 29 (5) | 20 (22) | 32 (20) | 25 (11) | 16 (3)
  Interproximal: Day 34 | 23 (21) | 54 (10) | 22 (11) | 27 (18) | 19 (14) | 34 (30) | 37 (19) | 36 (25) | 25 (15) | 14 (9) | 10 (7) | 27 (14) | 23 (11) | 25 (3)
  Facial: Eligibility | 15 (14) | 35 (36) | 22 (11) | 17 (10) | 11 (7) | 29 (4) | 24 (11) | 35 (21) | 22 (14) | 17 (3) | 16 (13) | 17 (13) | 10 (11) | 10 (11)
  Facial: Day 0 | 16 (9) | 39 (39) | 28 (13) | 16 (5) | 10 (7) | 20 (4) | 22 (16) | 35 (28) | 31 (17) | 11 (5) | 25 (19) | 25 (14) | 22 (18) | 12 (7)
  Facial: Day 14 | 16 (13) | 37 (37) | 19 (11) | 29 (10) | 11 (10) | 17 (8) | 19 (13) | 34 (13) | 23 (18) | 19 (15) | 19 (10) | 29 (9) | 12 (8) | 11 (5)
  Facial: Day 28 | 12 (13) | 27 (34) | 22 (9) | 20 (16) | 5 (4) | 23 (15) | 23 (19) | 23 (10) | 23 (18) | 22 (5) | 13 (13) | 27 (28) | 16 (11) | 6 (0)
  Facial: Day 34 | 14 (16) | 46 (17) | 15 (9) | 15 (16) | 11 (7) | 21 (19) | 24 (13) | 27 (16) | 22 (19) | 10 (4) | 8 (4) | 22 (18) | 16 (12) | 18 (11)
  Lingual: Eligibility | 16 (18) | 18 (16) | 30 (12) | 26 (23) | 24 (27) | 26 (9) | 36 (19) | 38 (32) | 28 (8) | 17 (8) | 23 (19) | 21 (5) | 16 (9) | 13 (7)
  Lingual: Day 0 | 25 (19) | 34 (22) | 29 (15) | 23 (7) | 22 (16) | 33 (5) | 35 (23) | 41 (29) | 30 (14) | 27 (13) | 25 (20) | 30 (14) | 21 (14) | 22 (1)
  Lingual: Day 14 | 16 (18) | 19 (11) | 22 (13) | 20 (15) | 23 (21) | 14 (14) | 31 (22) | 33 (31) | 25 (13) | 21 (15) | 20 (9) | 35 (6) | 19 (8) | 19 (13)
  Lingual: Day 28 | 19 (23) | 21 (24) | 28 (13) | 27 (13) | 22 (17) | 27 (9) | 42 (26) | 33 (13) | 26 (15) | 25 (7) | 22 (23) | 35 (10) | 258 (8) | 20 (2)
  Lingual: Day 34 | 23 (21) | 45 (4) | 20 (15) | 28 (16) | 21 (20) | 36 (34) | 39 (22) | 36 (28) | 21 (8) | 13 (8) | 11 (8) | 27 (11) | 23 (10) | 21 (3)

ADVERSE EVENTS:
Time Frame: up to 28 days
Description: Formal statistical analysis of the safety data was not performed due to the small sample size.
Arm/Group | Phase 1, 1a (2mg) | Phase 1, 1a Placebo | Phase 1, 2a (4mg) | Phase 1, 2a Placebo | Phase 1, 3a (6mg) | Phase 1, 3a Placebo | Phase 1, 4a (10mg) | Phase 1, 4a Placebo | Phase 1, 5a (20mg) | Phase 1, 5a Placebo | Phase 1, 6a (30mg) | Phase 1, 6a Placebo | Phase 1, 7a (50mg) | Phase 1, 7a Placebo | Phase 1, 8a (75mg) | Phase 1, 8a Placebo | Phase 1, 9a (100mg) | Phase 1, 9a Placebo | Phase 2, 1b (4mg) | Phase 2, 1b Placebo | Phase 2, 2b (6mg) | Phase 2, 2b Placebo | Phase 2, 3b (10mg) | Phase 2, 3b Placebo | Phase 2, 4b (20mg) | Phase 2, 4b Placebo | Phase 2, 5b (30mg) | Phase 2, 5b Placebo | Phase 2, 6b (50mg) | Phase 2, 6b Placebo | Phase 2, 7b (75mg) | Phase 2, 7b Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/4 | 0/2 | 0/4 | 0/2 | 0/4 | 0/2 | 0/7 | 0/3 | 0/7 | 0/3 | 0/7 | 0/3 | 0/7 | 0/3 | 0/7 | 0/3 | 0/4 | 0/2 | 0/7 | 0/3 | 0/7 | 0/2 | 0/7 | 0/3 | 0/7 | 0/3 | 0/7 | 0/3 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/4 | 0/2 | 0/4 | 0/2 | 0/4 | 0/2 | 0/7 | 0/3 | 0/7 | 0/3 | 0/7 | 0/3 | 0/7 | 0/3 | 0/7 | 0/3 | 0/4 | 0/2 | 0/7 | 0/3 | 0/7 | 0/2 | 0/6 | 0/3 | 0/7 | 0/3 | 0/7 | 0/3 | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/4 | 0/2 | 0/4 | 1/2 | 0/4 | 1/2 | 1/7 | 2/3 | 0/7 | 0/3 | 0/7 | 0/3 | 2/7 | 0/3 | 2/7 | 0/3 | 2/4 | 1/2 | 3/7 | 1/3 | 3/7 | 0/2 | 1/6 | 2/3 | 5/7 | 2/3 | 5/7 | 1/3 | 5/7 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, 1a (2mg) (N=2) | Phase 1, 1a Placebo (N=1) | Phase 1, 2a (4mg) (N=4) | Phase 1, 2a Placebo (N=2) | Phase 1, 3a (6mg) (N=4) | Phase 1, 3a Placebo (N=2) | Phase 1, 4a (10mg) (N=4) | Phase 1, 4a Placebo (N=2) | Phase 1, 5a (20mg) (N=7) | Phase 1, 5a Placebo (N=3) | Phase 1, 6a (30mg) (N=7) | Phase 1, 6a Placebo (N=3) | Phase 1, 7a (50mg) (N=7) | Phase 1, 7a Placebo (N=3) | Phase 1, 8a (75mg) (N=7) | Phase 1, 8a Placebo (N=3) | Phase 1, 9a (100mg) (N=7) | Phase 1, 9a Placebo (N=3) | Phase 2, 1b (4mg) (N=4) | Phase 2, 1b Placebo (N=2) | Phase 2, 2b (6mg) (N=7) | Phase 2, 2b Placebo (N=3) | Phase 2, 3b (10mg) (N=7) | Phase 2, 3b Placebo (N=2) | Phase 2, 4b (20mg) (N=6) | Phase 2, 4b Placebo (N=3) | Phase 2, 5b (30mg) (N=7) | Phase 2, 5b Placebo (N=3) | Phase 2, 6b (50mg) (N=7) | Phase 2, 6b Placebo (N=3) | Phase 2, 7b (75mg) (N=7) | Phase 2, 7b Placebo (N=3)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation in throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose urine present (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coating in mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device connection issue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema, hard palate, right side, molar area (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdomin discomfort, upper stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oral mucosal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puffy and wrinkling sensation, bilateral buccal mucosa (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stiffness of neck and shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Teeth staining (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tongue pigmentation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothh discoloration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No